CLINICAL TRIAL: NCT07187765
Title: Respiratory Safety of Oliceridine in Propofol-Sedated Gastrointestinal Endoscopy: A Double-Blind, Randomized Controlled Trial
Brief Title: Respiratory Safety of Oliceridine During Sedated Gastrointestinal Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiyou Wei (Other)
Responsible Party: Sponsor-Investigator, Shiyou Wei, Department of Anesthesiology, Shanghai Pulmonary Hospital, Shanghai, China
Organization: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20250254
Record Dates: First submitted 2025-08-06; First posted 2025-09-23 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Hypoxemia During Surgery; Gastrointestinal Endoscopy
Keywords: Hypoxemia; Gastrointestinal Endoscopy; Oliceridine; Sufentanil; Deep Sedation
MeSH Terms: conditions — Hypoxia | interventions — ((3-methoxythiophen-2-yl)methyl)((2-(9-(pyridin-2-yl)-6-oxaspiro(4.5)decan-9-yl)ethyl))amine; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Both participants and investigators will be blinded to group allocation. Study medications (Oliceridine or Sufentanil) will be prepared in identical syringes by a nurse not involved in patient care or outcome assessment, ensuring that neither patients nor clinicians are aware of the treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oliceridine Group (Experimental): Patients in this group will receive intravenous oliceridine (1 mg for gastroscopy or 1.5 mg for colonoscopy) combined with propofol (1-2 mg/kg) for sedation during gastrointestinal endoscopy.
  Interventions: Drug: Oliceridine
- Sufentanil Group (Active Comparator): Patients in this group will receive intravenous sufentanil (5 μg for gastroscopy or 7.5 μg for colonoscopy) combined with propofol (1-2 mg/kg) for sedation during gastrointestinal endoscopy.
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Oliceridine — Oliceridine will be administered intravenously at a dose of 1 mg for gastroscopy or 1.5 mg for colonoscopy, in combination with propofol (1-2 mg/kg), to provide sedation and analgesia during gastrointestinal endoscopy.
  Other Names: TRV130
  Arms: Oliceridine Group
Drug: Sufentanil — Sufentanil will be administered intravenously at a dose of 5 μg for gastroscopy or 7.5 μg for colonoscopy, in combination with propofol (1-2 mg/kg), to provide sedation and analgesia during gastrointestinal endoscopy.
  Other Names: Sufentanil Citrate
  Arms: Sufentanil Group

SUMMARY:
This study is a prospective, single-center, double-blind, randomized controlled trial designed to evaluate the effect of oliceridine versus sufentanil on the incidence of hypoxemia in adult patients undergoing gastrointestinal endoscopy under deep sedation. The trial will compare the rates of hypoxemia (defined as SpO₂ ≤92%) between the two analgesic regimens when combined with propofol. The primary aim is to determine whether oliceridine can reduce the incidence of hypoxemia compared to sufentanil during endoscopic procedures.

DETAILED DESCRIPTION:
Gastrointestinal endoscopy is frequently performed under deep sedation to minimize patient discomfort caused by mechanical stimulation. Currently, the combination of propofol and short-acting opioids, such as sufentanil, is widely used for its reliable sedation and analgesia. However, opioid-induced respiratory depression (OIRD) remains a notable concern. Unlike traditional opioids, oliceridine is a synthetic μ-opioid receptor agonist that preferentially activates G protein pathways while substantially reducing β-arrestin pathway activation, which may lower the risk of opioid-related adverse events, including respiratory depression.

Previous studies suggest that oliceridine is as effective as morphine for pain control and may be associated with a lower incidence of adverse effects, particularly in elderly or obese surgical patients. Clinical data also suggest a lower risk of respiratory depression with oliceridine compared to traditional opioids, but the incidence of hypoxemia with oliceridine during real-world deep sedation remains unclear.

This study aims to enroll adult patients (aged ≥18 years, ASA I-III) scheduled for elective gastrointestinal endoscopy. Participants will be randomly assigned (1:1) to receive either oliceridine (1 mg for gastroscopy or 1.5 mg for colonoscopy) or sufentanil (5 μg for gastroscopy or 7.5 μg for colonoscopy), both in combination with propofol (1-2 mg/kg). The primary outcome is the incidence of SpO₂ ≤92% from the start of sedation to the end of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥ 18 years.
* Scheduled to undergo elective gastrointestinal endoscopy (gastroscopy or colonoscopy).
* American Society of Anesthesiologists (ASA) physical status I-III.
* No history of severe cardiopulmonary dysfunction or other major systemic disease.

Exclusion Criteria:

* Dementia or any cognitive impairment precluding provision of informed consent.
* Known contraindication to oliceridine.
* Chronic (long-term) opioid use.
* Any other medical or logistic condition that, in the investigator's judgment, makes the participant unsuitable for the study (specify reason).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2025-09-22 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Hypoxemia (SpO₂ ≤92%) During Sedation for Gastrointestinal Endoscopy | From the start of sedation to the end of the gastrointestinal endoscopic procedure (approximately 1-60 minutes)
  The proportion of participants who experience hypoxemia, defined as a peripheral oxygen saturation (SpO₂) ≤92%, at any time from the start of sedation until the end of the endoscopic procedure.

SECONDARY OUTCOMES:
Incidence of secondary hypoxemic events during sedation for gastrointestinal endoscopy | From the start of sedation to the end of the gastrointestinal endoscopic procedure (approximately 1-60 minutes)
  The proportion of participants who experience any of the following between the start of sedation and the end of the endoscopic procedure :
  1. Severe hypoxemia, defined as lowest SpO₂ ≤ 85%
  2. A drop in SpO₂ of > 5% relative to the participant's highest measured value during the sedation period

OTHER OUTCOMES:
Number of participants requiring hypoxemia rescue interventions | From the start of sedation to the end of the gastrointestinal endoscopic procedure (approximately 1-60 minutes)
  Number of participants who, during sedation, required one or more of the following airway/ventilatory rescue measures to treat hypoxemia: none, mask ventilation, jaw-thrust maneuver, tracheal intubation, or other.
Total propofol dose administered | From the start of sedation to the end of the gastrointestinal endoscopic procedure (approximately 1-60 minutes)
  Cumulative amount of propofol (in mg) administered intravenously to each participant for sedation during the endoscopic procedure.
Incidence of opioid-related adverse events within 1 hour post-procedure | 1 hour after endoscopic procedure
  Proportion of participants experiencing any of the following within the first hour after procedure completion: nausea, vomiting, hypoxemia, pruritus, or dizziness.
Incidence of intra-procedural anesthesia-related adverse events | From initiation of sedation to completion of endoscopic procedure
  Proportion of participants who, during sedation, experienced any of: procedure interruption due to anesthesia (e.g. patient movement, hypoxemia), bradycardia, tachycardia, hypotension, hypertension, or required administration of vasoactive medications (vasopressors or chronotropes).

CONTACTS AND LOCATIONS:
Overall Officials: Shiyou Wei, PhD, Study Chair — 上海市肺科医院
Locations (1):
- Tianmen First People's Hospital, Tianmen, Hubei, China

IPD SHARING:
Plan to Share IPD: No